CLINICAL TRIAL: NCT06551831
Title: End-of-life Decision-making Among Young Patients With Advanced Cancer: a Grounded Theory Approach
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202406142RINE
Record Dates: First submitted 2024-08-04; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: End-of-life Decision-making
Keywords: Young Patients; Advanced Cancer; Grounded Theory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young Patients With Advanced Cancer: 1. The patient has a solid tumor.
  2. The age at initial cancer diagnosis is between 15 and 39 years.
  3. The patient is at least 18 years old at the time of enrollment.
  4. The patient has cancer with metastasis, either present at initial diagnosis or occurring after treatment or follow-up.
  5. After metastasis, the first-line curative treatment is ineffective.

SUMMARY:
The purpose of this qualitative research is to use grounded theory to explore and describe the thoughts of young advanced cancer patients regarding end-of-life care and how these thoughts influence the related decision-making process.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a solid tumor.
* The age at initial cancer diagnosis is between 15 and 39 years.
* The patient is at least 18 years old at the time of enrollment.
* The patient has cancer with metastasis, either present at initial diagnosis or occurring after treatment or follow-up.
* After metastasis, the first-line curative treatment is ineffective.

Exclusion Criteria:

- Patients who, for any reason, including severe psychological distress (as determined by the attending physician, psychiatrist, or specialist nurse based on assessments and impressions during routine patient care), cognitive impairment, or physical limitations (such as frailty), are unable to communicate or participate in an interview lasting more than 30 minutes.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: * The patient has a solid tumor.
  * The age at initial cancer diagnosis is between 15 and 39 years.
  * The patient is at least 18 years old at the time of enrollment.
  * The patient has cancer with metastasis, either present at initial diagnosis or occurring after treatment or follow-up.
  * After metastasis, the first-line curative treatment is ineffective.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Interview Guide | 2024/7~2025/7
  1.The journey since diagnosis. 2. The most profound or recent medical decision. 3. The most profound or recent medical decision. 4. Anticipated future medical decisions. 5. Future end-of-life care options

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No